CLINICAL TRIAL: NCT00254254
Title: A Randomized, Single-Blind, Dose-Rising, Placebo-Controlled, Crossover Study to Evaluate the Pharmacokinetics, Pharmacodynamics, and Tolerability of Exenatide in Adolescent Subjects With Type 2 Diabetes Mellitus
Brief Title: A Study to Evaluate the Pharmacokinetics, Pharmacodynamics, and Tolerability of Exenatide in Adolescent Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2993-124
Record Dates: First submitted 2005-11-14; First posted 2005-11-16 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; adolescents; exenatide; Amylin; Lilly
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sequence 1 (Experimental): Exenatide 2.5 mcg - Exenatide 5 mcg - Placebo 0.02 mL
  Interventions: Drug: Exenatide - Exenatide - Placebo
- Sequence 2 (Experimental): Exenatide 2.5 mcg - Placebo 0.02 mL - Exenatide 5 mcg
  Interventions: Drug: Exenatide - Placebo - Exenatide
- Sequence 3 (Experimental): Placebo 0.02 mL - Exenatide 2.5 mcg - Exenatide 5 mcg
  Interventions: Drug: Placebo - Exenatide - Exenatide

INTERVENTIONS:
Drug: Exenatide - Exenatide - Placebo — Exenatide 2.5 mcg, single dose, followed by Exenatide 5 mcg, single dose, followed by placebo 0.02 mL, single dose. All are subcutaneous injections.
  Other Names: Byetta
  Arms: Sequence 1
Drug: Exenatide - Placebo - Exenatide — Exenatide 2.5 mcg, single dose, followed by placebo 0.02 mL, single dose, followed by Exenatide 5 mcg, single dose. All are subcutaneous injections.
  Other Names: Byetta
  Arms: Sequence 2
Drug: Placebo - Exenatide - Exenatide — Placebo 0.02 mL, single dose, followed by Exenatide 2.5 mcg, single dose, followed by Exenatide 5 mcg, single dose. All are subcutaneous injections.
  Other Names: Byetta
  Arms: Sequence 3

SUMMARY:
This study will be the first evaluation of exenatide in adolescent subjects with type 2 diabetes mellitus and is designed to evaluate the blood levels of the drug (pharmacokinetics), the drug's biochemical and physiological effects (pharmacodynamics), and tolerability of exenatide in these subjects.

ELIGIBILITY:
Inclusion Criteria:

* Treatment with diet and exercise alone or a stable dose of metformin, or sulfonylurea, or metformin plus a sulfonylurea for at least 3 months.
* Has HbA1c 6.0% to 11.0%, inclusive, at screening.
* Has a body weight of >= 50 kg at screening.

Exclusion Criteria:

* Received any investigational drug or has participated in any type of clinical trial within 3 months prior to screening.
* Currently participates in any other interventional study.
* Is currently treated with any of the following excluded medications:

  * Sulfonylurea chlorpropamide
  * Thiazolidinedione within 3 months of screening.
  * Αlpha glucosidase inhibitor within 3 months of screening.
  * Meglitinide within 3 months of screening.
  * Insulin within 3 months of screening.
  * Pramlintide within 3 months of screening.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2006-02; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
To assess the pharmacokinetics of exenatide | Three day-long (8 hour) assessments over a 5-week period
  To assess pharmacokinetics of exenatide by measuring peak plasma time, time to peak concentration, terminal elimination half-life, apparent elimination time constant, apparent clearance, apparent volume of distribution, and area under concentration curve.
To assess the pharmacodynamics of exenatide | Three day-long (8 hour) assessments over a 5-week period
  To assess the pharmacodynamics of exenatide by measuring plasma glucose, serum insulin, and plasma glucagon: absolute and incremental area under the curve 0-3 hours), absolute and incremental area under the curve (0-6 hours), areas under the concentration-time curve (0-6 h), peak plasma contration, and time to peak concentration.
Number of adverse events | Visit 2 through Visit 4
  Adverse events will be assessed at all visits after the Screening Visit [Visit 2 (first time subject is dosed) through Visit 4 (study termination)]. All events assessed with special attention to changes in vital signs, ECGs, and laboratory values

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Porter, MD, Study Director — Amylin Pharmaceuticals, LLC.
Locations (5):
- United States (5):
  - Research Site, Little Rock, Arkansas
  - Research Site, San Diego, California
  - Research Site, Denver, Colorado
  - Research Site, Louisville, Kentucky
  - Research Site, San Antonio, Texas

REFERENCES:
- [Derived] Malloy J, Capparelli E, Gottschalk M, Guan X, Kothare P, Fineman M. Pharmacology and tolerability of a single dose of exenatide in adolescent patients with type 2 diabetes mellitus being treated with metformin: a randomized, placebo-controlled, single-blind, dose-escalation, crossover study. Clin Ther. 2009 Apr;31(4):806-15. doi: 10.1016/j.clinthera.2009.04.005. PMID 19446153